CLINICAL TRIAL: NCT04958252
Title: Safety, Tolerability and Pharmacokinetics of Single Rising Oral Doses and Multiple Oral Doses of BI 1569912 in Healthy Male Japanese Subjects (Single-blind, Partially Randomised Within Dose Groups, Placebo-controlled, Parallel-group Design)
Brief Title: A Study in Healthy Japanese Men to Test How Different Doses of BI 1569912 Are Taken up by the Body and How Well They Are Tolerated
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1447-0004
Record Dates: First submitted 2021-07-06; First posted 2021-07-12 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Part A and Part B of the trial is designed as single-blind, partially randomised, and placebo-controlled within parallel dose groups.
  Part C is designed as a randomised, two-sequence, open-label, two period, two-way cross over trial.
Masking Description: Part A and Part B of the trial are designed single-blind (to participants). Part C is designed as open-label trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Part A: BI 1569912 low dose (Experimental)
  Interventions: Drug: BI 1569912
- Part A: BI 1569912 lower medium dose (Experimental)
  Interventions: Drug: BI 1569912
- Part A: BI 1569912 higher medium dose (Experimental)
  Interventions: Drug: BI 1569912
- Part A: BI 1569912 high dose (Experimental)
  Interventions: Drug: BI 1569912
- Part B: BI 1569912 low dose (Experimental)
  Interventions: Drug: BI 1569912
- Part B: BI 1569912 high dose (Experimental)
  Interventions: Drug: BI 1569912
- Part C: BI 1569912 (Experimental)
  Interventions: Drug: BI 1569912
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1569912 — BI 1569912
  Arms: Part A: BI 1569912 high dose; Part A: BI 1569912 higher medium dose; Part A: BI 1569912 low dose; Part A: BI 1569912 lower medium dose; Part B: BI 1569912 high dose; Part B: BI 1569912 low dose; Part C: BI 1569912
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The main objectives of this trial are to investigate safety and tolerability of BI 1569912 in healthy male Japanese subjects following oral administration of single rising doses and multiple doses.

Secondary objective is the exploration of pharmacokinetics (PK) of BI 1569912.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a medical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead Electrocardiogram (ECG), and clinical laboratory tests
* Japanese ethnicity, according to the following criteria: born in Japan, have lived outside of Japan <10 years, and have parents and grandparents who are Japanese
* Age of 18 to 45 years (inclusive)
* Body mass index (BMI) of 18.5 to 25.0 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation
* Subjects who agree to minimize the risk of making their partner pregnant by fulfilling any of the following criteria starting from the first administration of trial medication until 90 days after last administration of trial medication

  * Use of adequate contraception, any of the following methods plus condom: intrauterine device, combined oral contraceptives that started at least 2 months prior to the first drug administration.
  * Vasectomized (vasectomy at least 1 year prior to enrolment)
  * Surgical sterilization (including bilateral tubal occlusion, hysterectomy or bilateral oophorectomy) of the subject's female partner

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 40 to 90 mmHg, or pulse rate outside the range of 40 to 99 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-08-05 (Actual); Primary Completion 2023-10-24 (Estimated); Study Completion 2023-10-24 (Estimated)

PRIMARY OUTCOMES:
Part A and Part B: Percentage of subjects with drug-related adverse events | up to 27 days
Part C: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) | up to 3 days
Part C: Maximum measured concentration of the analyte in plasma (Cmax) | up to 3 days

SECONDARY OUTCOMES:
Part A: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 4 days
Part A: Maximum measured concentration of the analyte in plasma (Cmax) | up to 4 days
Part B, after the first dose: Area under the concentration-time curve of the analyte in plasma from 0 to 24 hours (AUC0-24) | up to 17 days
Part B, after the first dose: Maximum measured concentration of the analyte in plasma (Cmax) | up to 17 days
Part B, after the last dose: Area under the concentration-time curve of the analyte in plasma over the dosing interval τ at steady state (AUCτ,ss) | up to 17 days
Part B, after the last dose: Maximum measured concentration of the analyte in plasma at steady state (Cmax,ss) | up to 17 days
Part C: Percentage of subjects with drug-related adverse events | up to 3 days
Part C: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- SOUSEIKAI Sumida Hospital, Tokyo, Sumida-ku, Japan

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com